CLINICAL TRIAL: NCT02781818
Title: A Randomized, Controlled, Double-blind Study to Evaluate the Efficacy of Intralesional Triamcinolone in the Treatment of Hidradenitis Suppurativa.
Brief Title: A Randomized Controlled Trial Evaluating the Efficacy of Intralesional Triamcinolone in Hidradenitis Suppurativa.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-0773
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-02

CONDITIONS: Hidradenitis Suppurativa
Keywords: hidradenitis; intralesional; triamcinolone
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis | interventions — Triamcinolone Acetonide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Triamcinolone Acetonide 10mg/mL (Experimental): Each lesion randomized to this group will receive a single intralesional treatment with 0.1 mL of triamcinolone 10mg/mL solution.
  Interventions: Drug: Triamcinolone Acetonide 10mg/mL
- Triamcinolone Acetonide 40mg/mL (Experimental): Each lesion randomized to this group will receive a single intralesional treatment with 0.1 mL of triamcinolone 40mg/mL solution.
  Interventions: Drug: Triamcinolone Acetonide 40mg/mL
- Normal Saline Placebo (Placebo Comparator): Each lesion randomized to this group will receive a single intralesional treatment with 0.1 mL of sterile normal saline solution.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Triamcinolone Acetonide 10mg/mL — Triamcinolone acetonide is a glucocorticoid used in intralesional treatment of many skin diseases, intra-articular treatment of inflammatory joint diseases, and intramuscular treatment for systemic management of systemic inflammatory diseases. It is commonly used in clinical practice for the treatment of acute abscesses and nodules of hidradenitis suppurativa, but little clinical trial data exist supporting its use.
  Other Names: Kenalog®-10
  Arms: Triamcinolone Acetonide 10mg/mL
Drug: Triamcinolone Acetonide 40mg/mL — Triamcinolone acetonide is a glucocorticoid used in intralesional treatment of many skin diseases, intra-articular treatment of inflammatory joint diseases, and intramuscular treatment for systemic management of systemic inflammatory diseases. It is commonly used in clinical practice for the treatment of acute abscesses and nodules of hidradenitis suppurativa, but little clinical trial data exist supporting its use.
  Other Names: Kenalog®-40
  Arms: Triamcinolone Acetonide 40mg/mL
Drug: Normal Saline — Normal saline 0.1 mL will be administered intralesionally at the selected site.
  Other Names: Placebo
  Arms: Normal Saline Placebo

SUMMARY:
Purpose: To evaluate the effectiveness of intralesional triamcinolone for the treatment of hidradenitis suppurativa (HS)

Participants: Patients diagnosed with Hidradenitis Suppurativa that have active inflammatory HS lesions. Up to 60 lesions will be treated. Between 20 and 60 patients will be enrolled dependent on the number of lesions they have treated. (up to 3 per patient)

Procedures (methods): Injection of triamcinolone or placebo into active lesions of hidradenitis suppurativa

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled trial of two concentrations of intralesional triamcinolone, triamcinolone 40mg/mL and triamcinolone 10mg/mL, with normal saline as a placebo control. For subjects with lesions deemed appropriate for the study, between one and three treatment sites will be marked with sequential lettering with a skin marker and documented by body location. Baseline pain level of each lesion will be recorded. At that time each lesion will be randomized in a 1:1:1 fashion to be treated with intralesional triamcinolone 10mg/mL, triamcinolone 40mg/mL, or normal saline placebo.

Following treatment, subjects will be given a paper questionnaire that will ask them to rate their level of pain on a 1-10 scale for each lesion, and whether they believe the target lesion has resolved on days 1, 2, 3, 5, 7, 10, and 14. On day 14 they will also rate how helpful they think the treatment is on a scale of 0-4. These will be patient-reported outcomes only without any physician assessment as this is felt to be a more clinically relevant outcome.

Aim 1. Characterize and compare the 3 regimens in terms of days to resolution of treated lesion.

Hypotheses for Aim 1: Days to resolution of treated lesions will be fewer in the treatment groups compared to normal saline placebo, and will be fewer with triamcinolone 40mg/mL compared to triamcinolone 10mg/mL.

Aim 2. Characterize and compare the 3 regimens in terms of pain level on day 5.

Hypotheses for Aim 2: Rating of pain will be less in the treatment groups compared to normal saline placebo, and will be less with triamcinolone 40mg/mL compared to triamcinolone 10mg/mL at day 5.

Aim 3. Characterize and compare the 3 regimens in terms of patient rating of the "benefit of the treatment Hypotheses for Aim 1: Patient rating will be more favorable the treatment groups compared to normal saline placebo, and will be more favorable with triamcinolone 40mg/mL compared to triamcinolone 10mg/mL.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females > or = 16 years of age
2. Diagnosis or history of clinical features consistent with hidradenitis suppurativa for >1 year
3. Patient must have an inflammatory lesion at the time of treatment. This can be an inflammatory nodule defined by a tender, palpable subcutaneous nodule, or an abscess defined as as fluctuant, painful, subcutaneous nodule. Lesions greater than 2 centimeters in size will not be excluded. Inflammatory nodules or abscesses can be treated if they are associated with a sinus tract, which is a chronic HS lesion defined by tunneled lesion with multiple openings to the surface of the skin. Sinus tracts without associated nodules or abscesses will not be treatment targets.
4. Patient must be off of antibiotics or on a stable course of oral antibiotics for >4 weeks prior to the baseline visit. Allowable antibiotics during treatment course are topical clindamycin, topical chlorhexidine gluconate, oral doxycycline, oral minocycline, or oral clindamycin +/- rifampin.
5. Must be able to provide adequate informed consent for themselves

Exclusion Criteria:

1. Any patient with signs of active infection at the time of screening that is not related to their hidradenitis suppurativa
2. Patients who have been on non-permitted antibiotics in the 4 weeks prior to baseline. Allowable antibiotics during treatment course are topical clindamycin, topical chlorhexidine gluconate, oral doxycycline, oral minocycline, or oral clindamycin +/- rifampin.
3. Patients who have had surgical intervention of the treated body region (i.e., right axilla) beyond incision and drainage procedures in the last 8 weeks or with open surgical wounds in the treatment region.
4. Patients who have been started on immunomodulatory or biologic treatment (i.e., adalimumab, infliximab) in the past 4 weeks
5. Patients on non-stable doses of opiate analgesics for the last 14 days prior to screening
6. Patients with history of hypersensitivity reactions to triamcinolone
7. Ongoing health or physical exam concerns which the investigator feels may put the patient at significant risk

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Sayed, MD, Principal Investigator — UNC Dermatology; Erika Hanami, CCRC, Study Director — Project Manager
Locations (1):
- University of North Carolina Department of Dermatology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fajgenbaum K, Crouse L, Dong L, Zeng D, Sayed C. Intralesional Triamcinolone May Not Be Beneficial for Treating Acute Hidradenitis Suppurativa Lesions: A Double-Blind, Randomized, Placebo-Controlled Trial. Dermatol Surg. 2020 May;46(5):685-689. doi: 10.1097/DSS.0000000000002112. PMID 31490300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting to an academic dermatology department in a subspecialty hidradenitis suppurativa clinic were enrolled during clinic visits between 6/20/2016 and 5/17/2017
Pre-assignment Details: The design allows for individual subjects to have multiple lesions randomized to distinct treatment arms, which means a single subject could be included as participants in multiple arms. This results in the total participant number calculated by adding participants in each arm to be higher (55) than the number of subjects enrolled (32).
Units Other Than Participants: Lesions
Groups:
- Triamcinolone Acetonide 10mg/mL: Each lesion randomized to this group received a single intralesional treatment with 0.1 mL of triamcinolone 10mg/mL solution.
- Triamcinolone Acetonide 40mg/mL: Each lesion randomized to this group received a single intralesional treatment with 0.1 mL of triamcinolone 40mg/mL solution.
- Normal Saline Placebo: Each lesion randomized to this group received a single intralesional treatment with non-bacteriostatic 0.1 mL of sterile normal saline solution.
Period: Overall Study
Arm/Group | Triamcinolone Acetonide 10mg/mL | Triamcinolone Acetonide 40mg/mL | Normal Saline Placebo
Started | 20; 24 Lesions | 18; 22 Lesions | 17; 21 Lesions
Completed | 16; 18 Lesions | 16; 20 Lesions | 16; 20 Lesions
Not Completed | 4; 6 Lesions | 2; 2 Lesions | 1; 1 Lesions
Not completed — Lost to Follow-up | 4 | 2 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: lesions
Groups:
- Triamcinolone Acetonide 10mg/mL: Each lesion randomized to this group received a single intralesional treatment with 0.1mL of triamcinolone 10mg/mL solution.
- Triamcinolone Acetonide 40mg/mL: Each lesion randomized to this group received a single intralesional treatment with 0.1mL of triamcinolone 40mg/mL solution.
- Normal Saline Placebo: Each lesion randomized to this group received a single intralesional treatment with non-bacteriostatic 0.1mL of sterile normal saline solution.
- Total: Total of all reporting groups
Arm/Group | Triamcinolone Acetonide 10mg/mL | Triamcinolone Acetonide 40mg/mL | Normal Saline Placebo | Total
Number analyzed (Participants) | 16 | 16 | 16 | 48
Number analyzed (lesions) | 18 | 20 | 20 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 2
  Between 18 and 65 years | 15 | 15 | 14 | 44
  >=65 years | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 15 | 41
  Male | 4 | 2 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 6 | 8 | 23
  White | 7 | 10 | 8 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 16 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Days to Lesion Resolution in Combined Treatment Arms Compared to the Placebo Arm.
Description: Mean number of days that patient reports it takes for a lesion to resolve. This is defined as a return of the skin to baseline in the treated area and an absence of pain.
Time Frame: 1-14 days
Measure: Mean (95% Confidence Interval); unit: Days
Units Other Than Participants: Lesions
Arm/Group | Triamcinolone Acetonide 10mg/mL | Triamcinolone Acetonide 40mg/mL | Normal Saline Placebo
Number analyzed (Participants) | 16 | 16 | 16
Number analyzed (Lesions) | 18 | 20 | 20
Days | 10.8 [8.2 to 13.4] | 10.9 [8.8 to 12.9] | 9.35 [6.9 to 11.9]
Statistical Analysis 1: Comparison: Triamcinolone Acetonide 10mg/mL vs Normal Saline Placebo; Test type: Superiority; p = 0.77, Mixed Models Analysis
Statistical Analysis 2: Comparison: Triamcinolone Acetonide 40mg/mL vs Normal Saline Placebo; Test type: Superiority; p = 0.46, Mixed Models Analysis

2. Secondary Outcome: Change in Pain From Baseline to Day 5
Description: Patients will rate pain on a scale of 1-10 (1 being no pain, 10 being the worst possible pain) at the baseline visit and on day 5. A secondary outcome will compare reduction in pain on day 5 in the combined treatment groups compared to the placebo group, and between the two treatment arms.
Time Frame: Baseline, Day 5
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Lesions
Arm/Group | Triamcinolone Acetonide 10mg/mL | Triamcinolone Acetonide 40mg/mL | Normal Saline Placebo
Number analyzed (Participants) | 16 | 16 | 16
Number analyzed (Lesions) | 18 | 20 | 20
units on a scale | 2 [.65 to 3.3] | 2.3 [1.1 to 3.5] | 2.6 [1.4 to 3.9]
Statistical Analysis 1: Comparison: Triamcinolone Acetonide 10mg/mL vs Normal Saline Placebo; Test type: Superiority; p = .65, Mixed Models Analysis
Statistical Analysis 2: Comparison: Triamcinolone Acetonide 40mg/mL vs Normal Saline Placebo; Test type: Superiority; p = 0.98, Mixed Models Analysis

3. Secondary Outcome: Patient Rating of Impression of Treatment at Day 14
Description: Patients will rate their impression of the treatment for each site as follows:
  0. Made it worse;
  1. Not helpful;
  2. A little bit helpful;
  3. Moderately helpful;
  4. Very helpful
  Comparison of rating of impression of treatment between the combined treatment groups and placebo will be performed. Similar comparison will be performed between the triamcinolone 10mg/ml and triamcinolone 40mg/ml treatment arms.
Time Frame: 14 days
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Lesions
Arm/Group | Triamcinolone Acetonide 10mg/mL | Triamcinolone Acetonide 40mg/mL | Normal Saline Placebo
Number analyzed (Participants) | 16 | 16 | 16
Number analyzed (Lesions) | 18 | 20 | 20
units on a scale | 2.5 [1.8 to 4.3] | 2.5 [1.9 to 4.4] | 2.4 [1.7 to 4.1]
Statistical Analysis 1: Comparison: Triamcinolone Acetonide 10mg/mL vs Normal Saline Placebo; Test type: Superiority; p = 0.50, Mixed Models Analysis
Statistical Analysis 2: Comparison: Triamcinolone Acetonide 40mg/mL vs Normal Saline Placebo; Test type: Superiority; p = 0.70, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 14 days
Description: Adverse event collections was done by phone on or about day 14 following the study intervention.
Groups:
- Triamcinolone Acetonide 10mg/mL: Each lesion randomized to this group will receive a single intralesional treatment with 0.1mL of triamcinolone 10mg/mL solution.
  Triamcinolone Acetonide 10mg/mL: Triamcinolone acetonide is a glucocorticoid used in intralesional treatment of many skin diseases, intra-articular treatment of inflammatory joint diseases, and intramuscular treatment for systemic management of systemic inflammatory diseases. It is commonly used in clinical practice for the treatment of acute abscesses and nodules of hidradenitis suppurativa, but little clinical trial data exist supporting its use.
- Triamcinolone Acetonide 40mg/mL: Each lesion randomized to this group will receive a single intralesional treatment with 0.1mL of triamcinolone 40mg/mL solution.
  Triamcinolone Acetonide 40mg/mL: Triamcinolone acetonide is a glucocorticoid used in intralesional treatment of many skin diseases, intra-articular treatment of inflammatory joint diseases, and intramuscular treatment for systemic management of systemic inflammatory diseases. It is commonly used in clinical practice for the treatment of acute abscesses and nodules of hidradenitis suppurativa, but little clinical trial data exist supporting its use.
- Normal Saline Placebo: Each lesion randomized to this group will receive a single intralesional treatment with 0.1mL of sterile normal saline solution.
  Normal Saline: Normal saline 0.1mL will be administered intralesionally at the selected site.
Arm/Group | Triamcinolone Acetonide 10mg/mL | Triamcinolone Acetonide 40mg/mL | Normal Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT02781818/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT02781818/SAP_001.pdf